CLINICAL TRIAL: NCT02440347
Title: Efficacy and Safety of Pulpal Anesthesia After Anterior and Middle Superior Alveolar (AMSA) Nerve Block Obtained by Articaine Computer-controlled and Conventional Delivery
Brief Title: Effects of Articaine Computer-controlled and Conventional Delivery for Anterior and Middle Superior Alveolar Nerve Block
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Bozidar Brkovic, DDS, MSc, PhD, Professor, DDS PhD Professor, University of Belgrade
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 36/5-2015; 175021 (Other Grant/Funding Number: Ministry of Education, Science and Technological Development)
Record Dates: First submitted 2015-04-23; First posted 2015-05-12 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Local Anesthesia
Keywords: local anesthesia; articaine; AMSA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Computer controlled anesthetic delivery by Anaeject (Experimental): Patients received single dose of 0.6 ml of 4% articaine with epinephrine (1:100.000) by computer controlled anesthetic delivery system (C-CLADS) for AMSA nerve block
  Interventions: Device: Computer controlled anesthetic delivery by Anaeject
- Conventional anesthetic delivery by carpule syringe (Active Comparator): Patients received single dose of 0.6 ml of 4% articaine with epinephrine (1:100.000) by conventional anesthetic delivery for AMSA nerve block
  Interventions: Device: Conventional anesthetic delivery by carpule syringe

INTERVENTIONS:
Device: Computer controlled anesthetic delivery by Anaeject — Single dose of 0.6ml 4% articaine with epinephrine (1:100.000) delivered by computer controlled local anesthetic delivery system (Anaeject).
  Arms: Computer controlled anesthetic delivery by Anaeject
Device: Conventional anesthetic delivery by carpule syringe — Single dose of 0.6ml 4% articaine with epinephrine (1:100.000) delivered by conventional syringe (carpule syringe).
  Arms: Conventional anesthetic delivery by carpule syringe

SUMMARY:
The purpose of this study was to investigate and compare pulpal anesthesia and cardiovascular parameters obtained with 0.6 ml of 4% articaine with epinephrine (1:100.000) for anterior and middle superior alveolar nerve (AMSA) block performed by standard and computer-controlled delivery in healthy volunteers.

DETAILED DESCRIPTION:
Traditionally, pulpal anesthesia is obtained by infiltration or mandibular nerve block. However, it is not always possible to achieve complete pulpal anesthesia with previously mentioned anesthetic techniques.

It is well documented that administration of 0,6-0,9 ml of anesthetic solution with palatal approach with anterior middle superior injection (AMSA) provided successful pulpal anesthesia from central incisor to second premolar. In addition, palatal soft tissues from midpalate to free gingiva and from central incisor to first molar are fully anesthetized with AMSA. The injection site is located at a point that bisects the maxillary first and second premolars, and midway between the crest of the free gingival margin and mid-palatine suture. The needle is orientated at a 45-degree angle with the bevel facing the palatal tissue. AMSA presents intraosseous anesthetic technique.

Traditionally, palatal injection administered with conventional syringe was described as very painful. On the other hand, computer controlled local anesthetic delivery system (CCLADS) has been recommended for AMSA as a system which allows slow administration of anesthetic solution, with constant pressure. It was shown that AMSA do not provide undesired buccal and upper lip anesthesia.

The AMSA technique has been recommended for proce¬dures ranging from operative restorations, crown preparation to scaling and root planning.

The aim of this study is to evaluate and compare parameters of pulpal anesthesia and cardiovascular function after AMSA injection of 4% articaine with epinephrine (1:100.000), delivered by conventional syringe or CCLADS. Study sample will comprise 30 healthy (ASA1) volunteers who will receive 0.6 ml 4% articaine with epinephrine (1:100.000) by conventional syringe, and after two-week washout period the same amount of local anesthetic by CCLADS. Parameters of pulpal and soft tissue anesthesia (onset and duration) for all maxillary teeth on the anesthetized side, as well as parameters of cardiovascular function (systolic blood pressure, diastolic blood pressure, heart rate) will be monitored and compared.

ELIGIBILITY:
Inclusion Criteria:

* ASA I
* full maxillary dental arch
* vital maxillary teeth without caries, restorations, periodontal disease or history of trauma

Exclusion Criteria:

* allergies to local anesthetic solution ingredients, food and drugs
* alcohol and drugs abuse
* heavy tobacco smoking

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Duration of pulpal anesthesia | up to 64 minutes from baseline
  Duration of pulpal maxillary anesthesia of all maxillary teeth in anesthetized side of upper jaw assessed by electrical pulp testing at 2-minute intervals.

SECONDARY OUTCOMES:
Onset of pulpal anesthesia | Up to 8 minutes
  Pulpal response to electrical pulp tester measured up to 8 minutes after injection
Width of anesthetic field marginal-superior | 5 minutes
  Width of area of soft tissue numbness measured 5 minutes after injection
Width of anesthetic field medial-lateral | 5 minutes
  Width of area of soft tissue numbness measured 5 minutes after injection
Duration of soft tissue anesthesia buccal | Up to 120 min
  Duration of soft tissue numbness followed up to 120 minutes after injection
Duration of soft tissue anesthesia palatal | Up to 120 minutes
  Duration of soft tissue numbness followed up to 120 minutes after injection
Systolic blood pressure at baseline | 0 minutes
  Systolic blood pressure before injection
Systolic blood pressure at 5 minutes | 0, 5 minutes
  Changes in systolic blood pressure from baseline at the time of injection delivery
Systolic blood pressure at 10 minutes | 0, 10 minutes
  Changes in systolic blood pressure from baseline 5 minutes after injection delivery
Systolic blood pressure at 15 minutes | 0, 15 minutes
  Changes in systolic blood pressure from baseline 10 minutes after injection delivery
Systolic blood pressure at 20 minutes | 0, 20 minutes
  Changes in systolic blood pressure from baseline 15 minutes after injection delivery
Systolic blood pressure at 35 minutes | 0, 35 minutes
  Changes in systolic blood pressure from baseline 30 minutes after injection delivery
Diastolic blood pressure at baseline | 0 minutes
  Diastolic blood pressure before injection
Diastolic blood pressure at 5 minutes | 0, 5 minutes
  Changes in diastolic blood pressure from baseline at the time of injection delivery
Diastolic blood pressure at 10 minutes | 0, 10 minutes
  Changes in diastolic blood pressure from baseline 5 minutes after injection delivery
Diastolic blood pressure at 15 minutes | 0, 15 minutes
  Changes in diastolic blood pressure from baseline 10 minutes after injection delivery
Diastolic blood pressure at 20 minutes | 0, 20 minutes
  Changes in diastolic blood pressure from baseline 15 minutes after injection delivery
Diastolic blood pressure at 35 minutes | 0, 35 minutes
  Changes in diastolic blood pressure from baseline 30 minutes after injection delivery
Heart rate at baseline | 0 minutes
  Heart rate before injection delivery
Heart rate at 5 minutes | 0, 5 mninutes
  Changes in heart rate from baseline at the time of injection delivery
Heart rate at 10 minutes | 0, 10 minutes
  Changes in heart rate from baseline 5 minutes after injection delivery
Heart rate at 15 minutes | 0, 15 minutes
  Changes in heart rate from baseline 10 minutes after injection delivery
Heart rate at 20 minutes | 0, 20 minutes
  Changes in heart rate from baseline 15 minutes after injection delivery
Heart rate at 35 minutes | 0, 35 minutes
  Changes in heart rate from baseline 30 minutes after injection delivery

CONTACTS AND LOCATIONS:
Overall Officials: Bozidar M Brkovic, DDS, PhD, Principal Investigator — School of Dental Medicine, University of Belgrade; Dejan Cetkovic, DDS, Principal Investigator — School of Dental Medicine, University of Belgrade; Vladimir M Biocanin, DDS, PhD, Principal Investigator — Faculty of Pharmacy and Health, University of Travnik, Bosnia and Herzegovina; Marija S Milic, DDS, Principal Investigator — School of Dental Medicine, University of Belgrade; Ivana Brajic, DDS, Principal Investigator — School of Dental Medicine, University of Belgrade
Locations (1):
- School of Dental Medicine, University of Belgrade, Belgrade, Serbia